CLINICAL TRIAL: NCT00239525
Title: 3-D Transcranial Ultrasound Analysis Using Definity Injectable Suspension
Brief Title: 3-D Transcranial Ultrasound Analysis Study
Acronym: Definity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00008393
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Cerebrovascular Accident; Intracranial Hypertension
Keywords: Cerebrovascular Accident; Intracranial Hypertension
MeSH Terms: conditions — Stroke; Intracranial Hypertension | interventions — Injections; perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: 3-D ultrasound scanner — The availability of color flow Doppler combined with effective ultrasound contrast agents in transcranial sonography serves as a low cost, bedside method for evaluation and management of patients with cerebrovascular disease in spite of the image degrading properties of the skull.
Drug: Perflutren Protein-Type A Microspheres for injection — Activated DEFINITY® (Perflutren Lipid Microsphere) Injectable Suspension is indicated for use in patients with suboptimal echocardiograms to opacify the left ventricular chamber and to improve the delineation of the left ventricular endocardial border.Bolus: The recommended dose for activated DEFINITY® is 10 microliters (μL)/kg of the activated product by intravenous bolus injection within 30-60 seconds, followed by a 10 mL saline flush. If necessary, a second 10 microliters (μL)/kg dose followed by a second 10 mL saline flush may be administered 30 minutes after the first injection to prolong contrast enhancement. Infusion: The recommended dose for activated DEFINITY® is via an IV infusion of 1.3 mL added to 50 mL of preservative-free saline. The rate of infusion should be initiated at 4.0 mL/minute, but titrated as necessary to achieve optimal image enhancement, not to exceed 10 mL/minute.
  Other Names: Definity

SUMMARY:
The purpose of this study is to investigate real time 3-D ultrasound imaging of the brain for the diagnosis and evaluation of stroke.

DETAILED DESCRIPTION:
The objective of this proposal is to extend our previous advances to investigate real time 3-D ultrasound imaging of the brain for the diagnosis and evaluation of stroke. Over the last decade, with the availability of color flow Doppler combined with effective ultrasound contrast agents, a renaissance has occurred in transcranial sonography as a low cost, bedside method for evaluation and management of patients with cerebrovascular disease in spite of the image degrading properties of the skull. Our hypothesis is that we can combine new generations of 2D array transducers with ultrasound contrast agents and phase aberration correction to enable real time 3D ultrasound imaging and 3D color flow Doppler of the brain with a factor of 10 improvement in spatial resolution compared to conventional transcranial sonography for improved diagnosis and evaluation of stroke.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* persons <18 years old
* pregnant or nursing women
* history of neurological disease
* congenital heart defect
* severe liver dysfunction
* respiratory distress syndrome
* hypersensitivity or an allergic reaction to blood products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Phase aberration correction of skull bone | 6 months
  This study will look to improve adaptive signal processing techniques for phase aberration correction of the skull while incorporating ultrasound contrast agent to increase signal to noise ratio in an ultrasound B-scan system with high speed RF data acquisition and 2-D arrays.In addition,we hope to develop adaptive transcranial real time 3D ultrasound and real time 3D color flow Doppler scanning of the brain incorporating ultrasound contrast agent to increase signal to noise ratio. A clinical evaluation of adaptive transcranial ultrasound imaging of the brain with phase aberration correction and ultrasound contrast agent will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Laskowitz, MD, Principal Investigator — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Lindsey BD, Light ED, Nicoletto HA, Bennett ER, Laskowitz DT, Smith SW. The ultrasound brain helmet: new transducers and volume registration for in vivo simultaneous multi-transducer 3-D transcranial imaging. IEEE Trans Ultrason Ferroelectr Freq Control. 2011 Jun;58(6):1189-202. doi: 10.1109/TUFFC.2011.1929. PMID 21693401
- [Result] Ivancevich NM, Pinton GF, Nicoletto HA, Bennett E, Laskowitz DT, Smith SW. Real-time 3-D contrast-enhanced transcranial ultrasound and aberration correction. Ultrasound Med Biol. 2008 Sep;34(9):1387-95. doi: 10.1016/j.ultrasmedbio.2008.01.015. Epub 2008 Apr 18. PMID 18395321
- [Result] Smith SW, Ivancevich NM, Lindsey BD, Whitman J, Light E, Fronheiser M, Nicoletto HA, Laskowitz DT. The ultrasound brain helmet: feasibility study of multiple simultaneous 3D scans of cerebral vasculature. Ultrasound Med Biol. 2009 Feb;35(2):329-38. doi: 10.1016/j.ultrasmedbio.2008.08.016. Epub 2008 Oct 23. PMID 18947918